CLINICAL TRIAL: NCT00532805
Title: QUANTitative Chest Computed Tomography UnMasking Emphysema Progression in Alpha-1 Antitrypsin Deficiency
Brief Title: The Use of High Resolution Chest Computed Tomography in Alpha-1 Antitrypsin Deficiency
Acronym: QUANTUM-1
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); Alpha-1 Foundation (Other)
Responsible Party: Principal Investigator, Charlie Strange, Professor of Pulmonary Medicine, Medical University of South Carolina
Other Study IDs: RDCRN 5701; 1U54RR019498-01 (NIH)
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Alpha-1 Antitrypsin Deficiency
Keywords: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 50 cc of serum at visits baseline, 6 months, 12 months, 18 months, 24 months and 36 months will be retained. These are kept at the University of Florida in the laboratory of Dr. Mark Brantly.
  There is an associated but independent DNA collection that is done if the patient is willing through an independent study and consent process with the University of Florida Alpha-1 DNA and Tissue Bank. This is a public resource with a scientific advisory committee with samples available for researcher access.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Individuals with a deficiency of alpha-1 antitrypsin (AAT) often develop emphysema. Traditional lung function tests may not be the most accurate way to measure the progression of emphysema. This study will compare high resolution computed tomography (CT) scans to spirometry to measure the progression of emphysema.

DETAILED DESCRIPTION:
AAT deficiency is a genetic disorder associated with emphysema. Spirometry, the lung function test that measures how well the lungs exhale air, is used to diagnose and track the progression of emphysema. Some studies have suggested that forced expiratory volume in 1 second (FEV1) measurements, a type of spirometry test, may lack accuracy in detecting disease progression in cases of severe AAT deficiency. Another method, high resolution chest CT scans, may be more accurate at measuring the progression of emphysema. The purpose of this study is to determine if high resolution CT scans are better at detecting the progression of emphysema than lung function tests. Results from this study may lead to the development of a more accurate way to assess lung tissue loss and may improve the understanding of lung destruction in AAT deficiency.

This study will last 4 years and will enroll people with AAT deficiency who have nearly normal lung function test results. Study visits, each lasting about 4 hours, will occur at baseline and months 6, 12, 18, 24, and 36. At each visit, participants will undergo lung function tests, a CT scan, blood collection, and a physical exam. Female participants will have urine collected for a pregnancy test. All participants will also complete questionnaires to assess health status and lung function. Study researchers will call participants every 2 months to collect information on lung disease symptoms and medication changes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AAT deficiency, as determined by both of the following conditions:

  1. Serum A1-P1 levels less than 11uM or 80 mg/dL
  2. Protease inhibitor phenotype Z (PiZZ) or Znull phenotype confirmed by gene probe analysis. Previous serum levels and phenotype results are acceptable if documented from a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory.
* FEV1 greater than or equal to 80% of the predicted value

Exclusion Criteria:

* Pregnant or intending to become pregnant within 4 years of study entry
* Previous lung transplantation
* Sibling of a participant who is already enrolled in the study
* Unable to attend scheduled clinic visits
* Currently smokes cigarettes or marijuana or quit smoking cigarettes or marijuana in the 1 year prior to study entry
* Current or planned use of oral tobacco products or nicotine replacement products
* Evidence of significant long-term or acute inflammation outside the lung, including connective diseases, panniculitis, or acute infection
* Unwilling to alter bronchodilator medications for 24 hours prior to scheduled quantitative CT (QCT) scans
* Musculoskeletal disease that limits exercise by walking
* Required to take any of the following medications within 48 hours of scheduled lung function testing: dicyclomine (Bentyl), propantheline (Pro-Banthine), mepenzolate (Cantil), methscopolamine (Pamine), and scopolamine (Transderm-Scop)
* Known allergy or intolerance to tiotropium or albuterol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with alpha-1 antitrypsin who have nearly normal lung function tests. Participants will be identified from patients of the investigators, physician referral, and the Alpha-1 Foundation Research Registry.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2007-08; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
CT density slope | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Strange, MD, Study Chair — Medical University of South Carolina
Locations (7):
- United States (7):
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Florida Medical Center, Gainesville, Florida
  - Harvard/Brigham and Women's Hospital, Boston, Massachusetts
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina